CLINICAL TRIAL: NCT05056974
Title: A Phase II Proof-of-concept Trial to Evaluate the Safety and Efficacy of UB-421 Plus Chidamide in Changing HIV Reservoirs Among ART Stabilized HIV-1 Patients Who Undergo ART Interruption
Brief Title: A Proof-of-concept Trial to Evaluate the Safety and Efficacy of UB-421 Plus Chidamide in Changing HIV Reservoirs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: United BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UBP-A232-HIV
Record Dates: First submitted 2021-08-18; First posted 2021-09-27 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2022-08

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — UB-421; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UB-421 + chidamide (Experimental): UB-421 + chidamide combination therapy
  Interventions: Biological: UB-421; Drug: chidamide

INTERVENTIONS:
Biological: UB-421 — 10 mg/kg, weekly UB-421 during the 8-week
Drug: chidamide — 10 mg/dose, twice a week for 8 weeks

SUMMARY:
This is a phase II proof-of-concept trial study to assess the safety and efficacy of UB-421 monotherapy plus chidamide in changing the latent HIV reservoir among ART-treated HIV-1 adults with stably viral suppression who undergo ART interruption.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 sero-positive, with documented HIV-1 infection by official, signed, written history
2. Male with body weight ≥ 50 kg or female with body weight ≥ 45 kg, aged 20 years or older.
3. No breastfeeding or pregnancy for women.
4. Have been receiving ART for more than 3 years by screening visit 1 (SV1).
5. Both male and female patients and their partners of childbearing potential must agree to use 2 medically accepted methods of contraception
6. Subjects must sign the informed consent before undergoing any study procedures.

Exclusion Criteria:

1. Subjects with active systemic infections, except for HIV-1
2. Any exposure to a monoclonal antibody within 12 weeks prior to the first dose of study drug.
3. Current receiving treatment regimen for hepatitis B, hepatitis C or latent tuberculosis
4. Any alcohol or illicit drug use
5. Receipt of any other investigational study agent(s) within 90 days before SV2.
6. Currently on the treatment for diabetes.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
HIV cell-associated RNA levels | Post-treatment weeks up to 48 weeks
  The change in HIV-1 Total DNA from baseline after study drug administration.

SECONDARY OUTCOMES:
HIV-1 Total DNA levels | Post-treatment weeks up to 48 weeks
  The changes in HIV-1 Total DNA levels during the study

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan, Taiwan